CLINICAL TRIAL: NCT01325441
Title: A Phase Ib/II Clinical Study of BBI608 Administered With Paclitaxel in Adult Patients With Advanced Malignancies
Brief Title: A Study of BBI608 Administered With Paclitaxel in Adult Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-201
Record Dates: First submitted 2011-03-25; First posted 2011-03-29 (Estimated); Results first posted 2023-02-03 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Cancer
Keywords: BBI608, thymic cancer
MeSH Terms: conditions — Neoplasms; Thymus Neoplasms | interventions — napabucasin; Paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- BBI608 and Paclitaxel 200mg BID (Experimental): Patients will receive BBI608 orally continuously at 200mg BID. A treatment cycle will be 4 weeks (28 days). BBI608 will be administered twice daily. On days 3, 10, and 17 of each 28 day cycle, patients will receive a 1 hour infusion of paclitaxel. Cycles will be repeated until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, adjustment is permitted.
  Interventions: Drug: BBI608; Drug: Paclitaxel
- BBI608 and Paclitaxel 240mg BID (Experimental): Patients will receive BBI608 orally continuously at 240mg BID. A treatment cycle will be 4 weeks (28 days). BBI608 will be administered twice daily. On days 3, 10, and 17 of each 28 day cycle, patients will receive a 1 hour infusion of paclitaxel. Cycles will be repeated until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, adjustment is permitted.
  Interventions: Drug: BBI608; Drug: Paclitaxel
- BBI608 and Paclitaxel 400mg BID (Experimental): Patients will receive BBI608 orally continuously at 400mg BID. A treatment cycle will be 4 weeks (28 days). BBI608 will be administered twice daily. On days 3, 10, and 17 of each 28 day cycle, patients will receive a 1 hour infusion of paclitaxel. Cycles will be repeated until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, adjustment is permitted.
  Interventions: Drug: BBI608; Drug: Paclitaxel
- BBI608 and Paclitaxel 480mg BID (Experimental): Patients will receive BBI608 orally continuously at 480mg BID. A treatment cycle will be 4 weeks (28 days). BBI608 will be administered twice daily. On days 3, 10, and 17 of each 28 day cycle, patients will receive a 1 hour infusion of paclitaxel. Cycles will be repeated until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, adjustment is permitted.
  Interventions: Drug: BBI608; Drug: Paclitaxel
- BBI608 and Paclitaxel 500mg BID (Experimental): Patients will receive BBI608 orally continuously at 500mg BID. A treatment cycle will be 4 weeks (28 days). BBI608 will be administered twice daily. On days 3, 10, and 17 of each 28 day cycle, patients will receive a 1 hour infusion of paclitaxel. Cycles will be repeated until progression of disease, unacceptable toxicity, or another discontinuation criterion is met. In the case of toxicity, adjustment is permitted.
  Interventions: Drug: BBI608; Drug: Paclitaxel

INTERVENTIONS:
Drug: BBI608
  Other Names: Napabucasin; BB608; BBI-608
Drug: Paclitaxel
  Other Names: Abraxane

SUMMARY:
This is an open label, single arm phase 1 dose escalation study and phase 2 study of BBI608 in combination with paclitaxel in patients with advanced malignancies.

DETAILED DESCRIPTION:
This is an open label, multi-center, single arm phase 1 dose escalation study and phase 2 study of BBI608 in combination with paclitaxel in patients with advanced solid tumors for whom weekly paclitaxel is an acceptable option.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent must be obtained and documented according to International Conference on Harmonization (ICH)- Good Clinical Practice (GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPPA) prior to study-specific screening procedures
2. A histologically or cytologically confirmed ovarian, breast, non-small cell lung, melanoma, gastric/GEJ/esophageal or other type of advanced cancer that is metastatic, unresectable, or recurrent and for which weekly paclitaxel is an acceptable therapeutic option.
3. Patients with epithelial ovarian, fallopian tube, or primary peritoneal cancer must also meet the following criteria: a. Must be either platinum-resistant or platinum-refractory according to the following definitions:(1)Platinum-resistant: a response to platinum therapy followed by progression within 6 months after completing therapy (2)Platinum-refractory: best response of stable disease or progression during platinum therapy; b. Must have had prior systemic treatment with a taxane; c. Must have received no more than 4 prior systemic cytotoxic regimens
4. Patients with melanoma must also meet the following criteria: a. If melanoma is BRAF wild-type or has BRAF mutations that are not amenable to BRAF inhibitor therapy, and the patient is a candidate for immunotherapy, must have received ipilimumab; b. If melanoma is positive for the V600E or V600K BRAF mutation, must have received at least one line of prior therapy with a BRAF-specific inhibitor; either alone or in combination.
5. Patients with triple negative breast cancer (estrogen receptor-negative (ER-), progesterone receptor-negative (PR-), and human epidermal growth factor receptor 2-negative (Her2-) must also meet the following criteria: a. Must have received at least one prior chemotherapy regimen for locally advanced or metastatic disease; b. Must have received prior taxane therapy.
6. Patients with NSCLC (adenocarcinoma, squamous, or adenosquamous histopathology) must also meet the following criteria: a. Must have disease that is stage IIIB, not curable by surgery or radiotherapy, or stage IV; b. Must have received at least one prior chemotherapy regimen for locally advanced or metastatic disease; c. EGFR-positive or ALK-positive patients must have received at least one line of EGFR-directed or ALK-directed therapy, respectively; d. Must have received prior taxane therapy.
7. Patients with adenocarcinoma arising from the esophagus, gastroesophageal junction, or stomach must also meet the following criteria: a. Must have received prior treatment with a platinum/fluoropyrimidine-based therapy with or without an anthracycline in the metastatic setting; or, in the adjuvant setting if recurrence occurred within 6 months of completing systemic adjuvant treatment; b. Patients with HER2 positive tumors must have had prior treatment with a Her2 inhibitor (e.g. trastuzumab or lapatinib); c. Patients who have received prior taxane therapy may be enrolled.
8. Patients with thymic carcinoma must have received at least one prior systemic chemotherapy regiment for metastatic, recurrent, locally advanced or otherwise unresectable disease.
9. ≥ 18 years of age
10. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1, see Section 9)
11. Karnofsky performance Status ≥ 70% (Section 15)
12. Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI608 dose
13. Females of childbearing potential must have a negative serum pregnancy test
14. Aspartate transaminase (AST) and alanine transaminase (ALT) £1.5 × upper limit of normal (ULN), or ≤ 2.5 × ULN with metastatic liver disease
15. Hemoglobin (Hgb) ≥ 10 g/dl
16. Total bilirubin £ 1.5 × ULN
17. Creatinine £ 1.5 ´ ULN or creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
18. Absolute neutrophil count ³ 1.5 x 109/L
19. Platelets ≥ 100 x 109/L
20. Life expectancy ≥ 3 months

Exclusion Criteria:

1. Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within 7 days of first dose provided all treatment-related adverse events have resolved or have been deemed irreversible, with the exception for a single dose radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 7 days before beginning the administration of BBI608.
2. Surgery within 4 weeks prior to first dose
3. Any known symptomatic brain metastases requiring steroids. Patients with treated brain metastases must be stable for 4 weeks after completion of that treatment, with image documentation required. Patients must have no clinical symptoms from brain metastases and must be either off steroids or on a stable dose of steroids for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated
4. Pregnant or breastfeeding
5. Significant gastrointestinal disorder(s), in the opinion of the Principal Investigator, (e.g., Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection)
6. Unable or unwilling to swallow BBI608 capsules daily
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements
8. Known severe hypersensitivity to paclitaxel
9. Abnormal ECGs (ie, QT prolongation - QTc > 480 msec, signs of cardiac enlargement or hypertrophy, bundle branch block, signs of ischemia or necrosis and Wolff Parkinson White patterns)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2011-04; Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lebedinsky, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (22):
- United States (17):
  - USC - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health (formerly Institute for Translational Oncology Research), Greenville, South Carolina
  - University of Tennessee Medical Center Cancer Institute, Knoxville, Tennessee
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology- Fort Worth, Fort Worth, Texas
  - Texas Oncology- Tyler, Tyler, Texas
  - Virginia Cancer Specialists, P.C., Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Compass Oncology- Northwest Cancer Specialists, Vancouver, Washington
- Canada (5):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - St. Mary's Hospital, Montreal, Quebec
  - McGill University Health Center-Glenn Site, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 565 participants were enrolled between April 2011 and March 2020.
Pre-assignment Details: Participants who died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Napabucasin 200mg BID Plus Paclitaxel: Participants received napabucasin 200mg administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 240mg BID Plus Paclitaxel: Participants received napabucasin 240mg administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 400mg BID Plus Paclitaxel: Participants received napabucasin 400mg administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 480mg BID Plus Paclitaxel: Participants received napabucasin 480mg administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 500mg BID Plus Paclitaxel: Participants received napabucasin 500mg administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
Period: Overall Study
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel
Started | 2 | 185 | 4 | 317 | 57
Completed | 2 | 185 | 4 | 317 | 57
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Napabucasin 200mg BID Plus Paclitaxel: Participants received napabucasin 200mg BID administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 240mg BID Plus Paclitaxel: Participants received napabucasin 240mg BID administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 400mg BID Plus Paclitaxel: Participants received napabucasin 400mg BID administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 480mg BID Plus Paclitaxel: Participants received napabucasin 480mg BID administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Napabucasin 500mg BID Plus Paclitaxel: Participants received napabucasin 500mg BID administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
- Total: Total of all reporting groups
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel | Total
Number analyzed (Participants) | 2 | 185 | 4 | 317 | 57 | 565
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (19.80) | 61.3 (10.14) | 64.8 (8.06) | 62.7 (10.42) | 60.5 (10.72) | 62.0 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 115 | 1 | 174 | 24 | 316
  Male | 0 | 70 | 3 | 143 | 33 | 249
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 149 | 4 | 259 | 49 | 463
  Hispanic | 0 | 9 | 0 | 11 | 0 | 20
  Black | 0 | 10 | 0 | 21 | 6 | 37
  Asian | 0 | 14 | 0 | 18 | 2 | 34
  Other | 0 | 3 | 0 | 8 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Assessment of safety of napabucasin administered in participants with advanced malignancies for whom weekly paclitaxel was an acceptable option by reporting of adverse events and serious adverse events
Time Frame: The time from the date of first treatment, while the patient is taking napabucasin, and for 30 days after stopping therapy, an average of 4 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel
Number analyzed (Participants) | 2 | 185 | 4 | 317 | 57
Participants | 2 | 183 | 4 | 317 | 57

2. Primary Outcome: Determination of the Recommended Phase 2 Dose by Assessing Dose-limiting Toxicities (DLTs)
Description: Determination of the Recommended Phase 2 dose (RP2D) of napabucasin when administered with paclitaxel in patients with advanced malignancies.
Time Frame: 28 days
Population: The Phase 1b portion of the study consisted of the first 24 patients enrolled in the study. These 24 patients, who received at least one dose of study drug, comprised the DLT Analysis Set.
Measure: Number; unit: mg
Groups:
- Napabucasin (BBI608) Plus Paclitaxel: All participants who were enrolled into the trial received napabucasin administered orally, twice daily, in combination with a fixed dose of paclitaxel administered IV weekly on day 3, 10 and 17 of each 28 day cycle.
Arm/Group | Napabucasin (BBI608) Plus Paclitaxel
Number analyzed (Participants) | 24
mg | 500

3. Secondary Outcome: Determination of the Maximum Observed Concentration (Cmax) and Area Under the Plasma Concentration vs. Time Curve (AUClast)
Description: To determine the maximum concentration of napabucasin and the area under the plasma concentration vs. time curve of napabucasin when administered in combination with weekly paclitaxel
Time Frame: Blood samples drawn on days 16 and 17 of the first study cycle
Population: Sponsor's decision to terminate further development of the napabucasin program. Data were not collected.
Arm/Group | Napabucasin (BBI608) Plus Paclitaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: Preliminary Anti-tumor Activity of BBI608 When Administered in Combination With Paclitaxel in Patients With Advanced Malignancies
Description: To assess the preliminary anti-tumor activity, specifically the objective response rate (ORR) of napabucasin administered in combination with paclitaxel. The Objective Response Rate (ORR) is the proportion of participants with a complete response or partial response who have measurable disease at baseline imaging.
Time Frame: From the date of first treatment, every 8 weeks, until the date of first documented objective disease progression, for an anticipated average of six months
Population: Data were not collected.
Arm/Group | Napabucasin (BBI608) Plus Paclitaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: The Objective Response Rate of Napabucasin Administered in Combination With Paclitaxel in Patients With Advanced Malignancies
Description: Assessment of the objective response rate (ORR) of napabucasin administered in combination with paclitaxel in patients with advanced malignancies.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; The Objective Response Rate (ORR) is the proportion of participants with a complete response or partial response.
Time Frame: From the date of first treatment, every 8 weeks, until the date of first documented objective disease progression, up to 60 months
Population: Patients had a baseline scan and at least 1 disease assessment following the initiation of therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel
Number analyzed (Participants) | 2 | 81 | 1 | 98 | 29
Participants | 0 | 23 | 0 | 9 | 6

6. Secondary Outcome: Disease Control Rate
Description: To determine the disease control rate (CDR) of napabucasin administered in combination with paclitaxel in patients with advanced malignancies.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. The Disease Control Rate (DCR) is the proportion of patients whose best overall response is CR, PR or SD.
Time Frame: as for outcome 5
Population: Patients who received at least 1 cycle of study treatment and had at least 1 disease assessment following the initiation of therapy. Patients missing imaging assessment following the initiation of treatment are not included in the assessment for DCR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel
Number analyzed (Participants) | 2 | 81 | 1 | 98 | 29
percentage of participants | 100 [15.8 to 100] | 53.1 [41.7 to 64.3] | 0 | 56.1 [45.7 to 66.1] | 51.7 [32.5 to 70.6]

7. Secondary Outcome: Progression Free Survival of Patients With Advanced Malignancies
Description: The effect of napabucasin given in combination with paclitaxel on Progression Free Survival (PFS) of patients with advanced malignancies.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: The time from the date of first treatment to the date of first documentation of disease progression or death due to any cause, up to 60 months
Population: Patients had a baseline scan and at least 1 on study scan or died from any cause.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel
Number analyzed (Participants) | 2 | 185 | 4 | 317 | 57
months | NA [NA to NA] — insufficient number of participants with events | 2.23 [1.87 to 3.52] | NA [NA to NA] — insufficient number of participants with events | 2.07 [1.87 to 2.53] | 2.3 [1.77 to 3.12]

8. Secondary Outcome: Overall Survival of Patients With Advanced Malignancies
Description: The effect of napabucasin given in combination with paclitaxel on Overall Survival (OS) of patients with advanced malignancies
Time Frame: 4 weeks after the patient has been off study treatment, every 3 months up to 18 months, then every 6 months thereafter until death, up to 118 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel
Number analyzed (Participants) | 2 | 185 | 4 | 317 | 57
months | NA [NA to NA] — insufficient number of participants with events | 7.79 [5.88 to 9.76] | NA [NA to NA] — insufficient number of participants with events | 6.51 [5.16 to 7.2] | 7.10 [3.75 to 9.07]

9. Secondary Outcome: Pharmacodynamics
Description: To determine the response (increase or decrease) of biomarkers from biopsied tumors following the administration of napabucasin
Time Frame: Day 17 of cycle 1
Population: No on-treatment biopsies were performed therefore no pharmacodynamic testing on tumor tissue was conducted.
Arm/Group | Napabucasin (BBI608) Plus Paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, up to 118 months.
Arm/Group | Napabucasin 200mg BID Plus Paclitaxel | Napabucasin 240mg BID Plus Paclitaxel | Napabucasin 400mg BID Plus Paclitaxel | Napabucasin 480mg BID Plus Paclitaxel | Napabucasin 500mg BID Plus Paclitaxel
All-Cause Mortality (participants affected / at risk) | 2/2 | 150/185 | 4/4 | 292/317 | 54/57
Serious Adverse Events (participants affected / at risk) | 1/2 | 15/185 | 2/4 | 28/317 | 7/57
Other Adverse Events (participants affected / at risk) | 2/2 | 183/185 | 4/4 | 317/317 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin 200mg BID Plus Paclitaxel (N=2) | Napabucasin 240mg BID Plus Paclitaxel (N=185) | Napabucasin 400mg BID Plus Paclitaxel (N=4) | Napabucasin 480mg BID Plus Paclitaxel (N=317) | Napabucasin 500mg BID Plus Paclitaxel (N=57)
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2 | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 5 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 3 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 1
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin 200mg BID Plus Paclitaxel (N=2) | Napabucasin 240mg BID Plus Paclitaxel (N=185) | Napabucasin 400mg BID Plus Paclitaxel (N=4) | Napabucasin 480mg BID Plus Paclitaxel (N=317) | Napabucasin 500mg BID Plus Paclitaxel (N=57)
Diarrhoea (Gastrointestinal disorders) | 2 | 137 | 4 | 268 | 49
Nausea (Gastrointestinal disorders) | 1 | 104 | 3 | 180 | 38
Abdominal pain (Gastrointestinal disorders) | 0 | 97 | 0 | 148 | 25
Vomiting (Gastrointestinal disorders) | 1 | 67 | 2 | 138 | 27
Abdominal distension (Gastrointestinal disorders) | 0 | 22 | 0 | 26 | 3
Flatulence (Gastrointestinal disorders) | 0 | 13 | 0 | 17 | 4
Fatigue (General disorders) | 2 | 107 | 3 | 189 | 36
Asthenia (General disorders) | 1 | 14 | 1 | 30 | 3
Oedema peripheral (General disorders) | 0 | 31 | 0 | 63 | 12
Decreased appetite (Metabolism and nutrition disorders) | 1 | 85 | 2 | 134 | 25
Dehydration (Metabolism and nutrition disorders) | 0 | 35 | 0 | 63 | 12
Hypokaelemia (Metabolism and nutrition disorders) | 0 | 28 | 0 | 58 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 15 | 0 | 50 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 47 | 0 | 123 | 20
Neutropenia (Blood and lymphatic system disorders) | 0 | 17 | 0 | 32 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 29 | 4
Neuropathy peripheral (Nervous system disorders) | 0 | 36 | 0 | 37 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 24 | 0 | 37 | 5
Dysgeusia (Nervous system disorders) | 0 | 11 | 0 | 16 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 64 | 0 | 73 | 17
White blood cell count decreased (Investigations) | 0 | 13 | 0 | 28 | 1
Weight decreased (Investigations) | 0 | 22 | 1 | 53 | 11
Neutrophil count decreased (Investigations) | 1 | 7 | 0 | 23 | 1
Chromaturia (Renal and urinary disorders) | 0 | 33 | 2 | 49 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 13 | 0 | 18 | 6
Constipation (Gastrointestinal disorders) | 1 | 41 | 0 | 50 | 12
Dysphagia (Gastrointestinal disorders) | 0 | 3 | 0 | 7 | 5
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 6 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 10 | 0 | 11 | 4
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 3
Pain (General disorders) | 0 | 6 | 0 | 14 | 6
Pyrexia (General disorders) | 1 | 26 | 1 | 48 | 6
Chills (General disorders) | 0 | 10 | 0 | 16 | 4
Disease progression (General disorders) | 0 | 10 | 0 | 18 | 4
Mucosal inflammation (General disorders) | 0 | 12 | 0 | 7 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 14 | 0 | 33 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 16 | 0 | 34 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 10 | 0 | 45 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 7 | 0 | 23 | 3
Headache (Nervous system disorders) | 0 | 27 | 0 | 20 | 8
Dizziness (Nervous system disorders) | 0 | 27 | 0 | 35 | 7
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 4
Paraesthesia (Nervous system disorders) | 0 | 7 | 0 | 7 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 52 | 1 | 73 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 43 | 0 | 44 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 27 | 1 | 28 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 8 | 0 | 22 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 22 | 2 | 20 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 17 | 0 | 25 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 4 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 8 | 0 | 9 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 18 | 0 | 11 | 6
Urinary tract infection (Infections and infestations) | 0 | 29 | 1 | 47 | 10
Candida infection (Infections and infestations) | 0 | 4 | 0 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 12 | 0 | 20 | 3
Proteinuria (Renal and urinary disorders) | 0 | 4 | 0 | 28 | 3
Insomnia (Psychiatric disorders) | 0 | 23 | 1 | 22 | 9
Confusional state (Psychiatric disorders) | 0 | 4 | 2 | 9 | 6
Depression (Psychiatric disorders) | 0 | 11 | 0 | 13 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 6 | 0 | 10 | 4
Hypotension (Vascular disorders) | 0 | 13 | 0 | 26 | 3
Influenza like illness (General disorders) | 1 | 3 | 0 | 9 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 7 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 14 | 0 | 58 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-05-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT01325441/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT01325441/SAP_001.pdf